CLINICAL TRIAL: NCT07167355
Title: Comparison of Outcome of Balloon Dilatation and Per Oral Endoscopic Myotomy in Children With Achalasia Cardia. A Randomized Control Cross Over Trial
Brief Title: Comparison of Balloon Dilatation and Per Oral Endoscopic Myotomy in Children With Achalasia Cardia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Director Interventional Endoscopy, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: COS 1
Record Dates: First submitted 2025-08-15; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Achalasia Cardia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POEM (Active Comparator)
  Interventions: Procedure: POEM
- BALLOON DILATATION (Active Comparator): Children randomised to BD arm, will undergo BD of 20mm (Controlled radial expansion [CRE], Boston Scientific) following an overnight fast. The balloon will be positioned at the gastroesophageal junction and inflated to a diameter of 20mm and a note will be made of whether the waist has disappeared or not. A repeat session of BD will be done after 1 month if TBE reveals a holdup of >5cm at 5 minutes. In this subgroup of children calculating Eckardt score will be difficult and unreliable.
  Balloon dilatation (children 7-17 years of age): Children randomised to BD arm will undergo BD of 30mm (Rigiflex II, Achalasia balloon dilators, Boston Scientific) following an overnight fast. The balloon will be positioned at the gastroesophageal junction and inflated to a diameter of 30mm with a pressure of 5psi initially and gradually the pressure will be increased to a maximum of 15 psi till the disappearance of waist fluoroscopically. A note will be made at the pressure at which the waist disappe
  Interventions: Procedure: BALLOON DILATATION

INTERVENTIONS:
Procedure: POEM — Children randomised to POEM arm will undergo a single session of POEM following an overnight fast. The procedure will be done in supine position under general anaesthesia. A gastroscope (Olympus GIF-HQ190) with a transparent tapered cap fit at its distal end will be used. A mucosal bleb will be created using a 21G sclerotherapy needle and a solution of saline with indigo-carmine dye. A posterior approach will be followed in all patients. A small mucosal incision (2-3mm) will be made using a needle knife and enlarged using an insulated tip knife (2-3cm). The submucosal tunned will then be entered and the submucosal fibres will be cleared using a triangular tip knife (TriangularTipKnife J, Olympus). Full thickness will be performed in all patients. Length of the myotomy will be ~3cm in the oesophagus and ~2cm in the cardia of the stomach. Minor bleeding will be controlled using coagulation forceps. Mucosal injury and resistance at the gastroesophageal junction will be examined. Mucosal i
  Arms: POEM
Procedure: BALLOON DILATATION — Children randomised to BD arm will undergo BD of 30mm (Rigiflex II, Achalasia balloon dilators, Boston Scientific) following an overnight fast. The balloon will be positioned at the gastroesophageal junction and inflated to a diameter of 30mm with a pressure of 5psi initially and gradually the pressure will be increased to a maximum of 15 psi till the disappearance of waist fluoroscopically. A note will be made at the pressure at which the waist disappears and will be maintained for 1 minute. One month after the initial session, if the Eckardt score >3 or if the TBE shows a barium column of >5cm at 5 minutes, a second session of BD will be done using a 35mm balloon.
  These children will be kept nil per oral for 4 hours post procedure. They will be observed for signs of perforation (crepitus, hemodynamic instability, chest pain). If they are stable, a clear liquid (water) will be provided. If there is no pain, they will be discharged with an advise to follow soft diet for a day
  Arms: BALLOON DILATATION

SUMMARY:
To compare the efficacy of balloon dilatation (BD) and per oral endoscopic myotomy (POEM) in improving the symptoms of children with achalasia in short and long term Presently most guidelines such as American Society for Gastrointestinal Endoscopy (ASGE) or European Society for Gastrointestinal Endoscopy (ESGE) recommend POEM or LHM or BD for the management of achalasia cardia based on the institutional expertise and patient preference. Only the Society of American Gastrointestinal and Endoscopic Surgeons (SAGES) recommend POEM or LHM over PBD for the management of achalasia in children. This is due to the lack of pediatric randomised control trial comparing the efficacy and safety of the two methods both in long and short term.

Children 3-18 years of age diagnosed as a case of achalasia cardia Place of trial: Department of medical gastroenterology, AIG Hospitals, Gachibowli and Somajiguda/Banjara Hills Duration of the trial: 3-4 years Sample size: 70 (35 each arm) Inclusion criteria: All children diagnosed as a case of achalasia cardia aged 3-18 years Exclusion criteria: Children who have undergone prior BD or POEM or Heller's myotomy. Type 3 achalasia cardia. Prior oesophageal/gastric surgery. Coagulopathy. Patients refusing consent for the trial.

Primary outcome: Percentage of children with achalasia cardia achieving a clinical success of BD and POEM at 12 months post intervention (clinical success is Eckardt score ≤ 3 and timed barium esophagogram (TBE) showing a holdup at gastroesophageal junction of <5cm at 5 minutes without requirement of further intervention) Secondary outcomes: Major and minor treatment complications, percentage patients developing gastroesophageal reflux disease, procedure time and improvement in growth Randomization: A stratified block randomization shall be performed using computer generated random number tables BD arm: Children <7 years of age will under 1-2 sessions of BD 1month apart with CRE 20mm balloon. Children 7-17 years of age will undergo 1-2 sessions of BD with Rigiflex II, Achalasia balloon dilator (30mm followed by 35mm).

POEM arm: Children 3-17 years of age will undergo 1 session of POEM as per the unit protocol.

Outcomes will be assessed at 3,6,12 months of the index procedure Crossover: If Eckardt score >3 and TBE showing a stasis of >5cm at 5 minutes, treatment is considered to have failed and crossover will be offered Endpoints: One year of follow up from the initial intervention or one year of follow up of the crossover intervention (in case of treatment failure), major complications.

Interim analysis: Following completion of follow up of 50% of the trial participants Early termination of trial: In case of any treatment modality having >10% major complications or during interim analysis one treatment modality significantly better than other (p<0.003)

DETAILED DESCRIPTION:
To compare the efficacy of balloon dilatation (BD) and per oral endoscopic myotomy (POEM) in improving the symptoms of children with achalasia in short and long term

Background:

Achalasia means "failure to relax". Achalasia cardia is a rare oesophageal motility disorder that occurs due to degeneration of the inhibitory myentric plexus of neurons of the oesophagus. This disorder is characterised by failure of relaxation of the lower oesophageal sphincter (LES), increased basal tone of the LES and absence of peristalsis in the oesophagus. All of these result in difficulty in passage of a food bolus from the oesophagus into stomach. Achalasia occurs in 0.1-0.18/100,000 per children per year.(1,2) Most patients present with symptoms of vomiting, dysphagia, chest pain and regurgitation. However, in children extra oesophageal symptoms such as chronic cough or aspiration is common. Smaller children may present with refusal to feed and failure to thrive. Achalasia cardia is a component of Allgrove syndrome and presents at an early age.(3) Treatment options for achalasia cardia include calcium channel blockers, botulinum injection, pneumatic balloon dilatation (BD), laparoscopic Hellers myotomy (LHM) and peroral endoscopic myotomy (POEM). BD, LHM and POEM are superior to the other therapies and should be offered to the patients when they are fit for the procedure. The type of achalasia, expertise of the centre and the patient preference should be taken into consideration before deciding on the modality of the treatment.(4) For type 3 achalasia cardia, POEM has been found to be superior when compared to BD or LHM.(4-7) However, for the other 2 types most guidelines don't provide a clear preference of one modality over the other. Major differences in the outcomes were not identified in between LHM and POEM in the systematic reviews and randomised control trials among type 1 and 2 achalasia.(8,9) Randomised control trials in adults have shown POEM to be superior to BD.(10,11) However, prospective comparative trials in children are lacking. A retrospective study by Tan Y et al showed BD to be as effective as POEM in short term (upto 1 year) but POEM was more effective on longer follow up.(12) Due to limited clinical trials and small sample sizes most guidelines advocate either of BD, LHM, POEM as the first line treatment modality for managing a patient with achalasia cardia on a case to case basis.(4-6) However, Society of American Gastrointestinal and Endoscopic Surgeons (SAGES) recommends for POEM or LHM as the preferred modality over BD even in type 1 and 2 achalasia cardia. SAGES guidelines though recognises the lack of pediatric randomised trials comparing the three modalities of treatment and recommends for comparative pediatric studies in the future.(7) BD is also not standardised in children and there is no recommendation on the size of balloon to be used at a particular age. Commonly most studies treat children more than 6 years of age similar to adults. There is a lack of clarity on the treatment of children below this age. Multiple studies have used different balloons of different sizes with varying success. The absence of standard Rigiflex balloon smaller than 30mm complicates the matter. POEM however, has been found to be safe in children and has been performed in smaller children with good success.(13-20) However, due to technical difficulty it is not yet being performed as a standard of care at all centres. Thus, with these deficiencies in the literature, we planned for a randomised control trial to compare the outcomes of BD and POEM in children.

Rationale Presently most guidelines such as American Society for Gastrointestinal Endoscopy (ASGE) or European Society for Gastrointestinal Endoscopy (ESGE) recommend POEM or LHM or BD for the management of achalasia cardia based on the institutional expertise and patient preference. Only the Society of American Gastrointestinal and Endoscopic Surgeons (SAGES) recommend POEM or LHM over PBD for the management of achalasia in children. This is due to the lack of paediatric randomised control trial comparing the efficacy and safety of the two methods both in long and short term.

Study participants Children 3-18 years of age diagnosed as a case of achalasia cardia Design: Randomized control crossover trial Place of trial: Department of medical gastroenterology, AIG Hospitals, Gachibowli and Somajiguda.

Duration of the trial: 3-4 years Sample size: 70 (35 each arm)

Randomization: A stratified block randomization shall be performed using computer generated random number tables BD arm: Children <7 years of age will under 1-2 sessions of BD 1month apart with CRE 20mm balloon. Children 7-17 years of age will undergo 1-2 sessions of BD with Rig flex II, Achalasia balloon dilator (30mm followed by 35mm).

POEM arm: Children 3-17 years of age will undergo 1 session of POEM as per the unit protocol.

Outcomes will be assessed at 3,6,12 months of the index procedure Crossover: If Eckardt score >3 and TBE showing a stasis of >5cm at 5 minutes, treatment is considered to have failed and crossover will be offered Endpoints: One year of follow up from the initial intervention or one year of follow up of the crossover intervention (in case of treatment failure), major complications.

Interim analysis: Following completion of follow up of 50% of the trial participants Early termination of trial: In case of any treatment modality having >10% major complications or during interim analysis one treatment modality significantly better than other (p<0.003)

ELIGIBILITY:
Inclusion Criteria:

-> All children of age 3-17 years diagnosed as a case of achalasia cardia

Exclusion Criteria:

* Children who had previously underwent BD, LHM or POEM
* Type 3 achalasia cardia. In children in whom HRM is not possible, if symptoms or barium oesophagogram is classical of type 3 achalasia, they will be excluded.
* Prior history of oesophageal or gastric surgery
* Coagulopathy
* Alternative diagnosis

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-09-03 (Estimated); Primary Completion 2027-10-22 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Primary: Clinical success is defined as • Eckardt score ≤ 3 • Absence of need for further endoscopic or surgical treatments to maintain Eckardt score ≤ 3 and • TBE showing oesophageal stasis of <5cm at 5minutes | 12 month
  • Eckardt score is calculated based on chest pain, regurgitation, dysphagia and weight loss

SECONDARY OUTCOMES:
Secondary objective: | 12 month
  • Major treatment related complications (treatment related complications were considered to be major if there was an unplanned hospital admission for > 24 hours, prolongation of a planned hospital admission, requirement of intensive care unit admission, requirement for a blood transfusion or need for additional endoscopic procedures for the management of the same)
Percentage of patients developing gastroesophageal reflux disease | 12 months
  Evidence of reflux esophagitis on upper gastrointestinal endoscopy
Minor complication rate | 12 months
  Number of patients developing minor complications (other than major complications)
Change in growth | 12 months
  improvement or worsening of growth following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Mohan Kumar Ramchandani, MD, DM, Principal Investigator — AIG Hospitals

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang X, Gong W, Deng Z, Zhou J, Ren Y, Zhang Q, Chen Z, Jiang B. Usefulness of peroral endoscopic myotomy for treating achalasia in children: experience from a single center. Pediatr Surg Int. 2015 Jul;31(7):633-8. doi: 10.1007/s00383-015-3717-9. Epub 2015 May 9. PMID 25957132
- [Background] de Moura ETH, Jukemura J, Ribeiro IB, Farias GFA, de Almeida Delgado AA, Coutinho LMA, de Moura DTH, Aissar Sallum RA, Nasi A, Sanchez-Luna SA, Sakai P, de Moura EGH. Peroral endoscopic myotomy vs laparoscopic myotomy and partial fundoplication for esophageal achalasia: A single-center randomized controlled trial. World J Gastroenterol. 2022 Sep 7;28(33):4875-4889. doi: 10.3748/wjg.v28.i33.4875. PMID 36156932
- [Background] Mayberry JF, Mayell MJ. Epidemiological study of achalasia in children. Gut. 1988 Jan;29(1):90-3. doi: 10.1136/gut.29.1.90. PMID 3343019